CLINICAL TRIAL: NCT05136222
Title: A Multi-centre Randomised Controlled Trial of Polysomnographic Titration of Non-invasive Ventilation in Motor Neurone Disease (PSG4NIVinMND; 3, Three Letter Acronyms [3TLA])
Brief Title: Polysomnographic Titration of Non-invasive Ventilation in Motor Neurone Disease
Acronym: 3TLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Austin Hospital, Melbourne Australia (Other); Institute for Breathing and Sleep, Australia (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other); Macquarie University, Australia (Other); Macquarie Health (Unknown); Western Sydney Local Health District (Other); Flinders Medical Centre (Other Government); Sir Charles Gairdner Hospital (Other); The Prince Charles Hospital (Other Government); Monash University (Other); Motor Neurone Disease Australia (Unknown); FightMND (Other); Australian Motor Neurone Disease Registry (Unknown); Calvary Bethlehem (Unknown); Perron Institute for Neurological and Translational Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT20020
Record Dates: First submitted 2021-10-21; First posted 2021-11-29 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Motor Neuron Disease / Amyotrophic Lateral Sclerosis
Keywords: Non-invasive ventilation; Polysomnography; Sleep study; Amyotrophic lateral sclerosis; Chronic respiratory failure
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with 12 month cohort follow-up
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The attending sleep scientist will refer to a database that reveals (statistician-generated) participant's treatment allocation. The sleep scientist will not reveal the treatment allocation to the Clinical team, Research team or the participant.
  Centralised allocation concealment will be ensured through the Adept/REDCap trial database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This trial of PSG-assisted commencement of non-invasive ventilation (NIV) in motor neurone disease (MND) follows the methodology of our previous single-site study (Hannan et al 2019 ERJ), with the addition of an open label cohort that extends until (the earlier of) 12 months or death.
  After empirical NIV set-up and an acclimatisation period (3 weeks), participants will undergo single night in-laboratory polysomnography (PSG). The PSG will be performed and supervised by a sleep scientist. In the intervention group, the "intervention" PSG results will be used to adjust/titrate NIV settings to optimize ventilation and improve synchrony between the patient and the NIV device. Participants will be asked to continue to use NIV as prescribed for the subsequent 7 week intervention period.
  Interventions: Other: Intervention polysomnography
- Control (Placebo Comparator): The participants allocated to the control group will also be asked to attend a single night in-laboratory PSG. The NIV settings will not be adjusted throughout the PSG ("sham" PSG). Participants in the control group will retain their original settings after the sham PSG, and will be asked to continue to use NIV in this manner for the subsequent 7 week intervention period.
  Interventions: Other: Sham polysomnography

INTERVENTIONS:
Other: Intervention polysomnography — Please refer to 'Arms: Intervention' section.
  Arms: Intervention
Other: Sham polysomnography — Please refer to 'Arms: Control' section.
  Arms: Control

SUMMARY:
A two-arm, individual participant randomised controlled, assessor-blinded trial in 7 MND care centres across Australia will be undertaken.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is a treatment that uses positive pressure delivered via a face mask or mouthpiece to assist a person to breathe. It can be used as a long-term treatment for people whose breathing is failing - usually due to chronic conditions that produce weakness of the respiratory muscles such as motor neurone disease / amyotrophic lateral sclerosis [MND/ALS]chronic obstructive pulmonary disease). Most people with MND/ALS use NIV at night initially. Even though NIV may improve survival and function, many are unable to use it for more than 4 hours per day (which is considered a threshold amount of use in order to gain a benefit) and many others are unable to tolerate it at all. Our team has recently provided evidence that specific and individualised titration of NIV leads to better outcomes in people with MND. This previous trial determined that the use of a sleep study (also called 'polysomnography') can improve the way people are initially set up with NIV. This study will replicate and extend the single site study in a large, multi-centre randomised controlled trial (RCT) across multiple sites This multi-centre RCT will also include a 12-month follow-up period to evaluate longer-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Clinical indication to commence long term NIV
* Confirmed clinical diagnosis of underlying condition

Exclusion Criteria:

* Medically unstable
* Hypoventilation attributable to medications with sedative/respiratory depressant side- effects
* Use of NIV for more than 1 month in the previous 3 months
* Inability to provide informed consent
* Previous intolerance of NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Adherence with NIV | Change during the acclimatization period (~3 weeks) and during the NIV treatment period (~7-8 weeks) (approx. 10 weeks total per participant).
  Defined as using NIV > 4 hours/day during the NIV treatment period.

SECONDARY OUTCOMES:
Intolerance of NIV | Change during the acclimatization period (~ 3 weeks) and during the NIV treatment period (~7-8 weeks) (approx. 10 weeks total per participant).
  Defined as cessation of NIV during the NIV treatment period and/or < 4 hours.
Respiratory function | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement as able.
  Forced expiratory volume in 1 second [FEV1], forced vital capacity [FVC]
Maximal inspiratory/expiratory pressure | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement as able.
  'MIPs/MEPs'.
Sniff nasal pressure | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement as able.
  'SNIP'.
Arousal index (during polysomnography) | During the baseline (following the ~3 week acclimatisation period) and during the follow-up assessment (~ week 3 + 7). Cohort: Not Collected.
  Defined as the number of electroencephalogram (EEG) arousals observed per hour of total sleep time (TST).
Asynchrony index (during polysomnography) | During the baseline (following the ~3 week acclimatisation period) and during the follow-up assessment (~ week 3 + 7). Cohort: Not Collected.
  Defined as the number of asynchrony events per hour of sleep.
Oxygen indices (during polysomnography) | During the baseline (following the ~3 week acclimatisation period) and during the follow-up assessment (~ week 3 + 7). Cohort: Not Collected.
  Multiple measures to summarise oxygenation as one single outcome including oxygen desaturation index (defined as the total number of oxygen desaturation episodes [= 4%] per hour of total), sleep time, nadir SpO2, and time with SpO2 < 90%, area under the curve and others.
Total sleep time (during polysomnography) | During the baseline (following the ~3 week acclimatisation period) and during the follow-up assessment (~ week 3 + 7). Cohort: Not Collected.
  Total amount of time asleep in minutes.
% rapid eye movement (REM) sleep (during polysomnography) | During the baseline (following the ~3 week acclimatisation period) and during the follow-up assessment (~ week 3 + 7). Cohort: Not Collected.
  Percentage of sleep characterised by eye movement, relaxation of the body, faster. respiration, and increased brain activity
% slow wave sleep (SWS) (during polysomnography) | During the baseline (following the ~3 week acclimatisation period) and during the follow-up assessment (~ week 3 + 7). Cohort: Not Collected.
  Percentage of 'deep sleep'.
Asynchrony sub-indices (during polysomnography) | During the baseline (following the ~3 week acclimatisation period) and during the follow-up assessment (~ week 3 + 7). Cohort: Not Collected.
  Ineffective efforts, double-trigger etc.
Dyspnoea Amyotrophic Lateral Sclerosis (DALS-15) | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement.
  A measure of breathlessness in people with ALS/MND.
Health-related quality of life - Severe Respiratory Insufficient Questionnaire (SRI) | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement.
  A measure of health-related quality of life.
Health-related quality of life - Assessment of Quality of Life (8-Dimension-AQoL) | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement.
  A measure of health-related quality of life.
Health-related quality of life - Calgary Sleep Apnoea Quality of Life Index (SAQLI) | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement.
  A measure of health-related quality of life.
Functional rating - Amyotrophic Lateral Sclerosis Functional Rating Scale (Revised) (ALSFRS) | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement.
  A clinical measure of functional rating in people with ALS/MND. Minimum score: 0, maximum score: 40. The higher the score the more function is retained.
Sleep quality - Pittsburgh Sleep Quality Index (PSQI) | RCT: During the baseline and during the follow-up assessment. Cohort: At 3, 6 and 12 months following RCT commencement.
  A measure of sleep quality.
Daytime somnolence - Epworth Sleepiness Scale (ESS) | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement.
  A measure of daytime sleepiness.
Daytime somnolence - Karolinska Sleepiness Scales (KSS) | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement.
  The KSS is rating of the current daytime sleepiness state using a 9-point scale (1 = very alert to 9 = very sleepy, fighting sleep).
Carer burden - Caregiver Burden Scale (CBS) | During the baseline (~week 0) and during the follow-up assessment (~ week 3 + 7). Cohort: At 3, 6 and 12 months following RCT commencement.
  A measure of caregiver burden. Rated ona scale from 0 (never) to 4 (nearly always), with higher scores indicating greater carer burden.
Cost effectiveness of the intervention | Throughout the trial period (approx. 5 years) (retrospective analysis).
  Economic evaluation using MBS/PBS data.
Usual clinical care practices | At trial commencement and trial end.
  Multidisciplinary clinician surveys at each recruitment site.
Usual care and the barriers and enablers to undertaking the intervention | At trial commencement (start of RCT) and trial end (end of RCT; approx. 4 to 5 years).
  Multidisciplinary clinician focus groups at each recruitment site.
Experience of receiving the intervention and the barriers and enablers to the PSG and NIV usage | At trial end (end of RCT; approx. 4 to 5 years)
  Participant semi-structured interviews.
Experience of the person they are caring for receiving the intervention and the barriers and enablers to the PSG and NIV usage | At trial end (end of RCT; approx. 4 to 5 years).
  Caregiver semi-structured interviews.

OTHER OUTCOMES:
Arterial Blood Gas (ABG) (during polysomnography) | RCT: During the baseline (following the acclimatisation period) and during the follow-up assessment. Cohort: Not Collected.
  Arterial Blood Gas

CONTACTS AND LOCATIONS:
Overall Officials: Abbey Sawyer, PhD, Study Chair — University of Melbourne
Locations (13):
- Australia (13):
  - Flinders Medical Centre, Adelaide
  - The Prince Charles Hospital, Brisbane
  - Motor Neurone Disease Australia, Canberra
  - Austin Health, Melbourne
  - Australian MND Registry, Melbourne
  - FightMND, Melbourne
  - Institute for Breathing and Sleep, Melbourne
  - Monash University, Melbourne
  - University of Melbourne, Melbourne
  - Sir Charles Gairdner Hospital, Perth
  - Macquarie University, Sydney
  - Royal Prince Alfred Hospital, Sydney
  - Westmead Hospital, Sydney

IPD SHARING:
Plan to Share IPD: Yes
Dataset in de-identified form will be shared on request to corresponding author.
Time Frame: 5 years from study completion.
Access Criteria: Subject to optional consent, where participants give permission for data to be used for the purpose of:
  1. The ethically approved research project only.
  2. This ethically approved research project and any closely related future research projects.
  3. This ethically approved research project and any future research projects that may or may not be related to this project.

REFERENCES:
- [Derived] Graco M, Berlowitz DJ, Sawyer A, Holland AE, Carey KA, Ahamed Y, Ridgers A, Lannin NA; 3TLA trial Group. Polysomnographic titration of non-invasive ventilation in motor neurone disease (3TLA): protocol for a process evaluation of a clinical trial. Trials. 2025 Mar 6;26(1):79. doi: 10.1186/s13063-025-08784-z. PMID 40050976
- [Derived] Berlowitz DJ, Rowe D, Howard ME, Piper A, Graco M, Braat S, Singh B, Souza TV, Lannin N, McLean A, Sawyer A, Carey KA, Ahamed Y; 3TLA Trial Group. Polysomnographic titration of non-invasive ventilation in motor neurone disease (3TLA): study protocol for a randomised controlled trial. Trials. 2025 Jan 6;26(1):10. doi: 10.1186/s13063-024-08464-4. PMID 39762986